CLINICAL TRIAL: NCT05430529
Title: Development and a Pilot Randomized Controlled Trial of a Brief Alcohol Intervention During Smoking Cessation Treatment Delivered by Healthcare Professionals
Brief Title: Alcohol Control in Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Derek Yee-Tak Cheung, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HKU_alcoholcontrol_protocol_v1
Record Dates: First submitted 2022-06-16; First posted 2022-06-24 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Smoking Cessation
Keywords: Alcohol Control; Intervention; Smoking Cessation; WhatsApp
MeSH Terms: conditions — Smoking Cessation | interventions — Control Groups; Ethanol; Methods

STUDY DESIGN:
Intervention Model Description: A 2-arm, parallel, single-blinded pilot randomized controlled trial to examine the feasibility, acceptability and potential efficacy of implementing the brief alcohol intervention in co-users of tobacco and alcohol.
Who Masked: Outcomes Assessor
Masking Description: All participants will be followed up via telephone by an allocation-blinded interviewer at 2-month after the random group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Alcohol Intervention for Intervention Group (Experimental): During the face-to-face smoking cessation counseling session, HCPs will first play a 2 - 3 minutes short video with electronic devices to participants who are allocated to intervention group.
  After the short video, HCPs will ask participants to share their thoughts and willingness of alcohol control. Participants are expected to show 4 responses: (1) refuse to attempt alcohol control; agree to attempt alcohol control that (2) quit drinking totally, (3) quit drinking for 2 weeks, or (4) reduce the alcohol consumption. HCPs will deliver personalized advice according to participants' choices and encourage them to receive the WhatsApp message reminders.
  In all participants, HCPs will invite them to receive WhatsApp messages reminders for incoming 4 weeks (3 messages per week).
  Nevertheless, HCPs can also choose to provide AUDIT-based brief intervention to the participants.
  Interventions: Behavioral: Standard Smoke Cessation Service; Behavioral: Brief Alcohol Intervention for Intervention Group
- Short Advice for Control Group (Active Comparator): If the control group participant encountering difficulties in smoke cessation caused by alcohol usage, HCP will provide short advice to them. Participant will be urged not to drink during smoke quitting. If drinking is unavoidable, participant should not drink exceed the low-risk drinking portion recommended by Department of Health, which is 2 standard alcohol units for men and 1 stand alcohol unit for women per day. HCPs will remind participants to aware their drinking portion, in order to quit smoke successfully.
  Interventions: Behavioral: Standard Smoke Cessation Service; Behavioral: Short Advice for Control Group

INTERVENTIONS:
Behavioral: Standard Smoke Cessation Service — Both of the intervention group and control group will receive standard smoke cessation service, which is same as usual practice.
Behavioral: Short Advice for Control Group — If the control group participant encountering difficulties in smoke cessation caused by alcohol usage, HCP will provide short advice to them. Participant will be urged not to drink during smoke quitting. If drinking is unavoidable, participant should not drink exceed the low-risk drinking portion recommended by Department of Health, which is 2 standard alcohol units for men and 1 stand alcohol unit for women per day. HCPs will remind participants to aware their drinking portion, in order to quit smoke successfully.
  Arms: Short Advice for Control Group
Behavioral: Brief Alcohol Intervention for Intervention Group — During the face-to-face smoking cessation counseling session, HCPs will first play a 2 - 3 minutes short video with electronic devices to participants who are allocated to the intervention group.
  After the short video, HCPs will ask participants to share their thoughts and willingness of alcohol control. Participants are expected to show 4 responses: (1) refuse to attempt alcohol control; agree to attempt alcohol control that (2) quit drinking totally, (3) quit drinking for 2 weeks, or (4) reduce the alcohol consumption. HCPs will deliver personalized advice according to participants' choices and encourage them to receive the WhatsApp message reminders.
  In all participants, HCPs will invite them to receive WhatsApp messages reminders for incoming 4 weeks (3 messages per week).
  In addition, HCPs can choose to discuss with participants the reasons for consuming alcohol.
  Nevertheless, HCPs can also choose to provide AUDIT-based brief intervention to the participants.
  Arms: Brief Alcohol Intervention for Intervention Group

SUMMARY:
This study aims to develop a theory-driven, brief alcohol intervention protocol for HCPs to deliver the intervention for co-users of tobacco and alcohol during smoking cessation treatment. The primary hypothesis is that smoking cessation treatment including the alcohol intervention will increase tobacco abstinence and reduce alcohol drinking. Our second hypothesis is that the brief intervention to deal with alcohol use will be feasible during smoking cessation treatment and be widely accepted by smokers.

DETAILED DESCRIPTION:
Co-use of Alcohol and Tobacco Co-use of tobacco and alcohol is common globally. Positive association of smoking and drinking at individual level has been found in both community settings and psychiatric epidemiological studies. In the U.S (2001-2002), about 21.7% of current drinkers were also current smokers, and about 34.8% of current smokers were current drinkers. In Hong Kong, according to the population-based study conducted by Hong Kong Council on Smoking and Health in 2018, about 22.2% and 9.3% of current smokers drank at least once a week and drank alcohol daily, respectively. From the client data (2014-16) of Tung Wah Group of Hospitals Integrated Centre on Smoking Cessation (TWGH-ICSC), the largest cessation service provider in Hong Kong, the prevalence of lower-risk drinking, increasing risk drinking, harmful drinking, and probable alcohol dependence, screened by the Alcohol Use Disorders Identification Test (AUDIT). in their clients is about 46.7%, 10.9%, 2.7% and 2.4%, respectively.

Co-use of tobacco and alcohol is harmful and incur substantial economic loss. Both tobacco and alcohol were classified by World Health Organization (WHO) as a Group 1 carcinogens. Concurrent use of tobacco and alcohol leads to 25.3% mortality due to coronary heart disease, stroke, respiratory and smoking-related cancer, compared with 20.5% among people who only smoked and 12.8% among who only had 15+ units of alcohol each week. Co-use of alcohol and tobacco also poses a severe economic burden on family and community. According to the Lancet's 2017 study, tobacco use costs global economies more than US$1 trillion annually through loss of productivity and health-care expenditure, while the weighted average cost of alcohol consumption ranged from 0.45 and 5.44% of Gross domestic Product (GDP)purchasing power parity (PPP) globally.

How Alcohol Use Hinders Smoking Cessation Alcohol consumption hinders smoking cessation, which can be explained by the theory in subjective reward effects, cross-substance cue reactivity, and other psychosocial factors. Based on the subjective reward effects, alcohol consumption increases nicotine's subjective rewarding effects, and hence increases satisfaction, liking, and calming feelings due to nicotine. Therefore, attempts to quit smoking are less successful among those with alcohol use disorder. The cross-substance cue reactivity suggested that there are cognitive or semantic associations between alcohol and cigarette use. That is, one substance will cue the use of the other substance. When alcohol and tobacco are used together for a number of times, the use of either substance will trigger a craving of another substance. This theory was commonly used to explain why alcohol is always an obstacle in smoking cessation and a cue for smoking relapse. These mechanisms have been supported by intervention trials and observational studies, showing that smoking rates among drinkers of different levels were significantly higher compared with non-drinkers after receiving smoking cessation treatment. If health care professionals (HCPs) do not handle smokers' drinking problems, they may miss the opportunity to help smokers to tackle the drinking problems at the same time.

Local Findings From the 2014-16 record of TWGH-ICSC, the self-reported quit rate at 26-week for clients with baseline AUDIT score 1-8, 9-15, and ≥16 after receiving the standard smoking cessation treatment was 43.4% (95% Confidence Interval (CI) 41.8%-45.1%), 37.1% (95%CI 33.8%-40.5%) and 26.7% (95%CI 22.4%-31.4%), respectively. The 52-week quit rate in these three drinking groups showed similar contrast (AUDIT score 1-8: 38.7%, 95%CI 37.0%-40.3%; 9-15: 31.9%, 95%CI 28.7%-35.2%; ≥16: 21.6%, 95%CI 17.7%-26.1%). Therefore, higher alcohol dependence is associated with lower abstinence in quit attempters who receive smoking cessation treatment. Two participants who self-reported tobacco abstinence for over a month from our ongoing qualitative study (funded by Health and Medical Research Fund (HMRF), ref no. 15163001) of smoking cessation stated that they were only smoking when they were drinking alcohol. They expressed that they smoked whenever they were drinking with friends and did not perceive occasional smoking during drinking episode as smoking relapse. All these results suggested that alcohol use reduces the effectiveness of smoking cessation treatment.

Interventions for Smoking and Drinking Co-use The above literature review suggested that a smoking cessation treatment that simultaneously addresses both alcohol and smoking problems is needed in clinical practice. The U.S. clinical practice guideline of treating tobacco use and dependence mentioned that helping smokers to recognize the dangerous situations of alcohol use is essential, and HCPs should instruct smokers to reduce/abstain from alcohol while quitting smoking. Previous study in alcohol treatment showed that alcohol users generally accept a concurrent treatment of both smoking cessation and alcohol.Combination of pharmacotherapy (i.e. varenicline and naltrexone) has been recommended to effectively and simultaneously treat heavy alcohol use and nicotine dependence.

Evidence-based brief intervention for reducing alcohol use has been established and is recommended by WHO. Behavioral interventions included personalized feedback, decisional balance, quit day setting and tailored skills-building. However, the effectiveness of these behavioral intervention for increasing tobacco abstinence and reducing alcohol use across the intervention trials is inconsistent. The investigators found 3 randomized controlled trials (RCTs) showed a promising effect of the intervention in increasing tobacco abstinence, but other 2 RCTs did not or even reduce tobacco abstinence rate. To late, there has been no systematic review on the effect of incorporating alcohol intervention into smoking cessation treatment. Therefore, the evidence is not yet conclusive.

Local Services for Alcohol Intervention Hospital Authority and non-governmental organizations are providing alcohol treatments, including Hospital Authority's Psychiatry Specialist Out-patient Clinics (SOPCs), Tung Wah Group of Hospitals Integrated Centre for Addiction Prevention and Treatment (ICAPT), TWGH's Alcohol Abuse Prevention and Treatment Service--"Stay Sober, Stay Free," and Alcoholics Anonymous Hong Kong. There has been no publication and data on the utilization of these services.

The Department of Health promoted screening and subsequently delivering a tailored health advice for alcohol users with AUDIT. It published a guide for HCPs to assess drinking and deliver an AUDIT-based brief alcohol intervention in primary health setting in 5-10 minutes. The first three questions of the AUDIT are grouped as AUDIT-C version, which attempts to quickly screen drinkers with high alcohol consumption level. If patients score 3 or above in AUDIT-C, HCPs will proceed to assess alcohol dependence with the rest of the AUDIT. The 3-rd question of the AUDIT-C ("How often do participants have at least 5 cans of beer/5 glasses of table wine/5 peg of spirits on one occasion?) is an indicator of binge-drinking.

According to the local guide on using AUDIT-based intervention, patients with lower-risk drinking (score 1-7in the AUDIT) should receive advice on health risks of drinking and they should drink less or abstain from alcohol. Patients with an increasing risk of drinking (score 8-15 in the AUDIT) should be warned on the increasing risk and impairment due to drinking, and they should cut down drinking. Patients with harmful drinking (score 16-19 in the AUDIT) usually have a pattern of alcohol use that is causing damage to health, hence they should receive a more severe warning and be encouraged to seek professional support. Patients who are defined as probable dependence (score 20 or above in the AUDIT) showed a cluster of behavioral, cognitive, and physiological phenomena, such as strong desire to consume alcohol, impaired self-control, persistent drinking, and physical withdrawal reaction). The HCPs should let them know that drinking is already causing alcohol dependence, and advise the patients to stop or reduce drinking under the help of professionals. It's best to refer patients in this category to a specialist for more in-depth evaluation and treatment. In addition to the above framework, pregnant women, persons on medication and persons with mental illnesses should be asked to abstain completely from alcohol.

Although this brief guide includes the instruction to educate drinkers the risks of excessive alcohol use and refer other services, there are several implementation difficulties. The guide was solely developed for alcohol reduction/abstinence, but it does not involve the intervention for alcohol and tobacco co-use. This guide does not address alcohol use as a barrier of quitting smoking. It does not instruct HCPs on aspects of beliefs, attitude and more personalized advice for smokers. The effectiveness and feasibility in adapting this AUDIT-based in clinical setting has not been evaluated. To address these limitations, an AUDIT-based brief alcohol intervention that can be specifically incorporated in smoking cessation treatment is needed. An alcohol intervention protocol customized for co-users, and training for HCPs about the knowledge, attitude, and practice of delivering alcohol and tobacco intervention are needed.

Proposed Alcohol Intervention In the proposed intervention, AUDIT will be tentatively adopted to screen potential participants. A need assessment will be done to guide the adaptation and revision of the final protocol. To increase the feasibility of applying the alcohol intervention, the need assessment is required to understand (1) current routine in smoking cessation treatment; (2) HCPs' capacity (knowledge, attitudes and practice) and acceptability of the intervention; (3) current co-users' expectations and acceptability of the intervention.

The aforementioned framework in delivering personalized advice to drinkers with lower-risk, drinking at increasing risk, harmful drinking and drinking dependence will be used. Co-users of tobacco and alcohol should be advised the importance of quitting smoking and reducing/abstaining alcohol. The investigators propose a short and brief interventions for co-users who are receiving smoking cessation treatment, because the investigators believe their primary goal is smoking cessation. The co-users may not have enough time or readiness to discuss the issue of drinking problems intensively. A brief advice on drinking may be more acceptable than an intensive intervention for these smokers.

The alcohol intervention protocol will be guided by the theory of self-determination and general health promotion action. The self-determination theory values the importance of internalized autonomy rather than external factors (e.g., requests from family members, friends, or healthcare professionals) during behavioral regulation. Previous RCT had revealed that participants who had the option to decide on their treatment showed a higher level of compliance with instructions. The positive association between autonomy and competence has also been shown by our previous RCT on smoking cessation. Compared with people with less autonomy in treatment, people with greater independence reported greater competence in achieving behavioral change.

The investigators' general health promotion action (GHPA) model stated that people with general intention to promote health are more likely to adopt specific health promotion actions. Specifically, smokers who have general intention to promote health are more likely to stop smoking. If co-users have the intention to improve health, they may pursue both alcohol reduction/abstinence and smoking cessation. One intervention RCT found that smokers who initiated a quit attempt could reduce alcohol consumption by 2.3 units per week after the target quit day, and heavier drinking smokers presented a more significant decrease (6.1 units) in alcohol intake. Based on this model, our proposed study shall encourage the HCPs to increase participants' awareness and intention for health and a healthy lifestyle.

Aims and Hypotheses to be Tested:

This study aims to develop a theory-driven, brief alcohol intervention protocol for HCPs to deliver the intervention for co-users of tobacco and alcohol during smoking cessation treatment. The primary hypothesis is that smoking cessation treatment including the alcohol intervention will increase tobacco abstinence and reduce alcohol drinking. Our second hypothesis is that the brief intervention to deal with alcohol use will be feasible during smoking cessation treatment and be widely accepted by smokers.

Setting The recruitment sites will be the smoking cessation clinics or services under TWGH-ICSC in Hong Kong, which offer behavioral and/or pharmacological interventions. The TWGH-ICSC operates 5 service centers, serving around 3000 smokers each year. The investigators have successful experience of collaborating with these service providers in recruiting smokers for several projects. For example, the investigators recruited around 1,000 smokers from these service providers in an HMRF-funded project in 2018-2019 (Project No. 15163001).

Procedures The HCPs who deliver the smoking cessation counselling will screen the eligibility of the clients at the first or later follow-up of their smoking cessation treatment, and invite eligible participants to join the RCT. When a counselor identifies a potential client, he/she will briefly introduce the alcohol control program. Participants who agree to join the RCT will be required to sign the consent form. HCPs will then randomize the client to either the intervention group or control group afterwards. In the intervention group, participants will receive the standard smoke cessation service and personalized advice on alcohol control. The details and key components of the intervention will be addressed in the intervention section below. In the control group, HCPs will deliver the standard smoke cessation service that same as the usual practice.

Randomization, Blinding The Qualtrics (an online platform for collecting data) randomizer function will be used for the randomization (with 1:1 allocation ratio) in this study. After participants consent to the study, HCPs will access Qualtrics for randomization. The Qualtrics will display the group allocation (either intervention group or control group) after HCPs enter the participants' names. HCPs will inform participants regarding their group allocation immediately. All HCPs and the participants will not be blinded to the given interventions. Outcome assessors at the telephone follow-up are blinded to the group allocation.

ELIGIBILITY:
Inclusion criteria:

* Self-report tobacco use in the past month
* Aged 18 or above
* Currently using or recently enrolled in local smoking cessation service
* Able to communicate in Cantonese/Mandarin and read Chinese
* Self-report alcohol use in either of the four drinking levels:
* Lower-risk of drinking problems (AUDIT score 1-7)
* Drinking at increasing risk (AUDIT score 8-15)
* Harmful drinking (AUDIT score 16-19)
* Having drinking dependence (AUDIT score >=20)
* Self-report one of the following:
* In previous quit attempts in lifetime, have smoked few cigarettes due to drinking alcohol (but not relapse)
* In the past 3 months, have felt an urge to smoking during/ after drinking
* In the past 3 months, smoked when drinking
* Smoked more cigarettes when drinking, compared to the day of smoke only
* In general, the drinking habit influenced the motivation to quit smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Self-reported Tobacco Abstinence in Past 7 Days | At 2 month follow-up.
  Number of Participants with Self-reported Tobacco Abstinence in Past 7 Days
Biochemically Validated tobacco abstinence at 2 month follow-up | At 2 month follow-up.
  Participants who report tobacco abstinence will be invited for a biochemical validation which defined participants as validated quitters if his/her exhaled carbon monoxide is 4ppm or below with a Bedfont Smokerlyzer or 30ng/ml below with the iScreen Oral Fluid Device (OFD) Cotinine Saliva Test Kit.
Alcohol consumption (alcohol units) in past week; | At 2 month follow-up.
  The alcohol consumption (alcohol units) in past week;
AUDIT score | At 2 month follow-up.
  The AUDIT score will be measured via the AUDIT questionnaire

OTHER OUTCOMES:
The feasibility of the intervention (intervention group only) | At 2 month follow-up.
  The feasibility will be assessed with the time required for the intervention and HCPs' compliance enquired in the action plan.
The acceptability of the intervention (intervention group only) | At 2 month follow-up.
  The acceptability will be assessed by the Treatment Acceptability/ Adherence Scale (TAAS) [24]. TAAS is a 7-point likert scale which ranged from 1 (disagree strongly) to 7 (agree strongly). It contains 11-item (e.g. ".The intervention is suitable for changing my drinking habits."). Higher score indicate higher degree of acceptability in this scale. Besides the TAAS, there are 6 additional open-ended questions will be used to collect participants' attitudes and feedback towards the intervention (e.g. "Please describe the most effective and unnecessary parts of the alcohol control brief intervention").

CONTACTS AND LOCATIONS:
Locations (1):
- Tung Wah Group of Hospitals Integrated Centre on Smoking Cessation, Hong Kong, Hong Kong

REFERENCES:
- [Background] Falk DE, Yi HY, Hiller-Sturmhofel S. An epidemiologic analysis of co-occurring alcohol and tobacco use and disorders: findings from the National Epidemiologic Survey on Alcohol and Related Conditions. Alcohol Res Health. 2006;29(3):162-71. PMID 17373404
- [Background] World Health Organization. AUDIT: The alcohol use disorders identification test: Guidelines for use in primary health care. World Health Organization; 2001.
- [Background] Hart CL, Davey Smith G, Gruer L, Watt GC. The combined effect of smoking tobacco and drinking alcohol on cause-specific mortality: a 30 year cohort study. BMC Public Health. 2010 Dec 24;10:789. doi: 10.1186/1471-2458-10-789. PMID 21184680
- [Background] The Lancet. Tobacco elimination: an economic and public health imperative. Lancet. 2017 Jan 21;389(10066):225. doi: 10.1016/S0140-6736(17)30132-0. Epub 2017 Jan 20. No abstract available. PMID 28118898
- [Background] Rose JE, Brauer LH, Behm FM, Cramblett M, Calkins K, Lawhon D. Potentiation of nicotine reward by alcohol. Alcohol Clin Exp Res. 2002 Dec;26(12):1930-1. doi: 10.1097/01.ALC.0000040982.92057.52. No abstract available. PMID 12500124
- [Background] Cook JW, Fucito LM, Piasecki TM, Piper ME, Schlam TR, Berg KM, Baker TB. Relations of alcohol consumption with smoking cessation milestones and tobacco dependence. J Consult Clin Psychol. 2012 Dec;80(6):1075-85. doi: 10.1037/a0029931. Epub 2012 Sep 10. PMID 22963593
- [Background] Rohsenow DJ, Monti PM, Colby SM, Gulliver SB, Sirota AD, Niaura RS, Abrams DB. Effects of alcohol cues on smoking urges and topography among alcoholic men. Alcohol Clin Exp Res. 1997 Feb;21(1):101-7. PMID 9046380
- [Background] Sayette MA, Martin CS, Wertz JM, Perrott MA, Peters AR. The effects of alcohol on cigarette craving in heavy smokers and tobacco chippers. Psychol Addict Behav. 2005 Sep;19(3):263-70. doi: 10.1037/0893-164X.19.3.263. PMID 16187804
- [Background] Fraser D, Kobinsky K, Smith SS, Kramer J, Theobald WE, Baker TB. Five population-based interventions for smoking cessation: a MOST trial. Transl Behav Med. 2014 Dec;4(4):382-90. doi: 10.1007/s13142-014-0278-8. PMID 25584087
- [Background] Leeman RF, McKee SA, Toll BA, Krishnan-Sarin S, Cooney JL, Makuch RW, O'Malley SS. Risk factors for treatment failure in smokers: relationship to alcohol use and to lifetime history of an alcohol use disorder. Nicotine Tob Res. 2008 Dec;10(12):1793-809. doi: 10.1080/14622200802443742. PMID 19023831
- [Background] Joseph AM, Nelson DB, Nugent SM, Willenbring ML. Timing of alcohol and smoking cessation (TASC): smoking among substance use patients screened and enrolled in a clinical trial. J Addict Dis. 2003;22(4):87-107. doi: 10.1300/j069v22n04_08. PMID 14723480
- [Background] Yardley MM, Mirbaba MM, Ray LA. Pharmacological Options for Smoking Cessation in Heavy-Drinking Smokers. CNS Drugs. 2015;29(10):833-45. doi: 10.1007/s40263-015-0284-5. PMID 26507831
- [Background] Beyer FR, Campbell F, Bertholet N, Daeppen JB, Saunders JB, Pienaar ED, Muirhead CR, Kaner EFS. The Cochrane 2018 Review on Brief Interventions in Primary Care for Hazardous and Harmful Alcohol Consumption: A Distillation for Clinicians and Policy Makers. Alcohol Alcohol. 2019 Jul 1;54(4):417-427. doi: 10.1093/alcalc/agz035. PMID 31062859
- [Background] Kahler CW, Metrik J, LaChance HR, Ramsey SE, Abrams DB, Monti PM, Brown RA. Addressing heavy drinking in smoking cessation treatment: a randomized clinical trial. J Consult Clin Psychol. 2008 Oct;76(5):852-62. doi: 10.1037/a0012717. PMID 18837602
- [Background] Toll BA, Martino S, O'Malley SS, Fucito LM, McKee SA, Kahler CW, Rojewski AM, Mahoney MC, Wu R, Celestino P, Seshadri S, Koutsky J, Hyland A, Cummings KM. A randomized trial for hazardous drinking and smoking cessation for callers to a quitline. J Consult Clin Psychol. 2015 Jun;83(3):445-54. doi: 10.1037/a0038183. Epub 2014 Nov 24. PMID 25419583
- [Background] Ames SC, Werch CE, Ames GE, Lange LJ, Schroeder DR, Hanson AC, Patten CA. Integrated smoking cessation and binge drinking intervention for young adults: a pilot investigation. Ann Behav Med. 2010 Dec;40(3):343-9. doi: 10.1007/s12160-010-9222-4. PMID 20730517
- [Background] Correa-Fernandez V, Diaz-Toro EC, Reitzel LR, Guo L, Chen M, Li Y, Calo WA, Shih YT, Wetter DW. Combined treatment for at-risk drinking and smoking cessation among Puerto Ricans: A randomized clinical trial. Addict Behav. 2017 Feb;65:185-192. doi: 10.1016/j.addbeh.2016.10.009. Epub 2016 Oct 22. PMID 27825036
- [Background] Pengpid S, Peltzer K, Puckpinyo A, Viripiromgool S, Thamma-Aphiphol K, Suthisukhon K, Dumee D, Kongtapan T. Screening and concurrent brief intervention of conjoint hazardous or harmful alcohol and tobacco use in hospital out-patients in Thailand: a randomized controlled trial. Subst Abuse Treat Prev Policy. 2015 May 27;10:22. doi: 10.1186/s13011-015-0018-1. PMID 26013537
- [Background] Centre for Health Protection, Department of Health. Alcohol Screening and Brief Intervention: A guide for use in primary care. 2017.
- [Background] Deci E, Ryan R. Handbook of Self-determination. Research. Rochester, NY: University of Rochester Press; 2002.
- [Background] Li WHC, Ho KY, Wang MP, Cheung DYT, Lam KKW, Xia W, Cheung KY, Wong CKH, Chan SSC, Lam TH. Effectiveness of a Brief Self-determination Theory-Based Smoking Cessation Intervention for Smokers at Emergency Departments in Hong Kong: A Randomized Clinical Trial. JAMA Intern Med. 2020 Feb 1;180(2):206-214. doi: 10.1001/jamainternmed.2019.5176. PMID 31790546
- [Background] Lam TH, Chan B, Ho SY, Chan WM. Stage of change for general health promotion action and health-related lifestyle practices in Chinese adults. Prev Med. 2004 Mar;38(3):302-8. doi: 10.1016/j.ypmed.2003.10.005. PMID 14766112
- [Background] Przulj D, Hajek P, Snuggs S, McRobbie H. Changes in Alcohol Consumption During a Stop-Smoking Attempt and Differences Between Smokers Using Nicotine Replacement and Smokers Using Varenicline. Nicotine Tob Res. 2018 Apr 2;20(5):583-588. doi: 10.1093/ntr/ntx105. PMID 28521015
- [Background] Milosevic I, Levy HC, Alcolado GM, Radomsky AS. The Treatment Acceptability/Adherence Scale: Moving Beyond the Assessment of Treatment Effectiveness. Cogn Behav Ther. 2015;44(6):456-69. doi: 10.1080/16506073.2015.1053407. Epub 2015 Jun 19. PMID 26091250
- [Background] Thorne S. Interpretive description. Developing qualitative inquiry. 2008.